CLINICAL TRIAL: NCT05748678
Title: A Study Evaluating the Efficacy of Cell-u-Light Apparel in Enhancing Lymph Drainage and Improving the Appearance of Grades of Cellulite in Affected Participants
Brief Title: Does Cell-U-Light Apparel Improve Cellulite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Whiteley Clinic (Other)
Collaborators: Canfield (Unknown)
Responsible Party: Principal Investigator, Mark Whiteley, Consultant Venous Surgeon, The Whiteley Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TWC-SM-2022-03
Record Dates: First submitted 2023-01-25; First posted 2023-03-01 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Cellulite
Keywords: compression; cellulite; appearance
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Intervention Model Description: Wearing apparell similar to cycling shorts which compresses the target area of the buttocks and thighs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of the compression apparel (Experimental): All participants
  Interventions: Device: Compression pants

INTERVENTIONS:
Device: Compression pants — Patients will have 3D photos taken each week of each buttock and thigh separately. A lymph scanner will also be used for each section to provide a percentage of water content. Weight will also be taken for each visit.
  The first 2 weeks the patients will wear their regular pants, and from weeks 3-7 wear the compression pants provided. Weeks 8-9 the patients will be asked to resume to regular pants again

SUMMARY:
This trial is arranged in 3 stages, lasting 8 weeks overall, designed to assess the before, during and after effects of the low-compression apparel with its integrated, variably raised, ink-polymer pads.

The study will recruit 21 (otherwise healthy) participants who are affected by cellulite. Volunteers will be selected in order to equally fill the 3 different grades of cellulite (7 volunteers of each grade (1, 2 & 3) - as Grade 0 is no evidence of cellulite, this category need not be included). Each volunteer will be 'sized' according to standard apparel sizing charts (as used by the manufacturer of the cycle shorts); Small (S), Medium (M), Large (L) and Extra Large (XL).

All participants will follow the same 3 stage sequence, which will involve a total of 9 short visits to The Whiteley Clinic, each lasting approximately 30 minutes. Upon completion of these visits, participants will each be offered £90 to subsidise their cost of travel - they will also be permitted to keep the low-compression apparel following the study. During each appointment, several measurements and assessment will be made:

* Standard demographics, weight, height, and any changes to dietary or exercise regimens over the trial period.
* Subjective assessment of the cellulite by the participant.
* Objective assessment and grading using the grading system described by Nunberger and Muller by the investigators
* Images of their cellulite-affected areas will be taken (this may include an area over the buttocks and an area over the thighs), using a high-resolution medical imaging (camera) system (Vectra H2 (https://www.canfieldsci.com/imaging-systems/vectra-h2-3d-imaging-system/)), to be independently assessed by Canfield Consultants and to be graded by a 'panel' of clinicians for objective classifications.
* Assessment of local lymphatic collections in the skin using a handheld lymph scanner to assess lymph accumulation (Delfin Lymphscanner, Delfin Technologies Ltd https://hadhealth.com/lymphscanner).
* During stage 2 only, participant assessment as to ease of donning and doffing the product, and comfort of wearing it.

DETAILED DESCRIPTION:
Stage 1:

The first stage of the trial is an induction and stabilisation phase. The participants will be seen on the first visit, the trail explained, and any questions answered. If the participant wishes to proceed, a consent form will be signed and the participant will be measured for the correct size Cell-u-Light product - but the product will NOT be given to the patient until visit 3, to prevent them from trying the product out before the trial stage.

They will then have the assessments performed and recorded. They will be given the time and dates of their next 8 weekly visits.

Visit 2 (end of week one) and visit 3 (end of week 3) will be part of stage 1. The Cell-u-light pants will not be given to the patient until visit 3 to

Stage 2:

The second stage of the trial will begin on the third visit (at the end of week 2) and will last for 4 weeks. Participants will be given the Cell-u-light low-compression apparel to wear and shown the correct method of donning and doffing. They will be instructed to wear them daily for a continuous 8-hour period. Participants can choose which 8 hours suits them best.

Participants will be instructed to remove the apparel a minimum of 2 hours before attending their appointments. This will allow time for small indentations left on the skin surface (caused by the ink-polymer pads) to dissipate, so that imaging and subjective assessments are accurate.

Stage 3:

The final stage will act as a 2 week 'wash-out' period. Participants will stop wearing the Cell-u-light and will have two final appointments at the clinic to record and observe any residual effects of the prior intervention.

Throughout the duration of the study, it will be vital that participants maintain their usual diet and exercise levels to avoid any fluctuations in weight (that may in turn affect the appearance of their cellulite). In this way, the investigators can ensure that any difference is due solely to the effects of Cell-u-Light. To further reduce deviations in weight, lymph abundance, etc. visits to the clinic will be standardised for each volunteer such that each appointment will be at the same time each week.

The trial will be performed in the clinical area in (the CQC registered) Whiteley Clinic. The temperature will be controlled and monitored to be within 20-22 centigrade. Consent for the trial and further usage of images in future publications will be obtained from all participants. [It will not be possible to ascertain which volunteer is being described from any photography.]

Participants will undergo non-invasive measurements, medical photographic imaging and scans to assess the following:

* Height - Only needed at the initial visit.
* Weight
* Appearance of cellulite
* Assessment of lymph in the thigh and buttock regions
* Subjective opinion of comfort and ease of donning and doffing of the apparel by participant
* Subjective grading of cellulite by participant
* Objective grading of cellulite by aesthetician

For the subjective grading of each participants' cellulite, the investigators will use the grading system described by Nunberger & Muller. This consists of 4 grades (0, 1, 2 and 3) as seen below, however, only 3 will be used as Grade 0 is the classification for 'no cellulite present' and therefore, does not fit the purpose of our study.

ELIGIBILITY:
Inclusion Criteria:

* Affected by stages 1, 2 or 3 of cellulite
* Can be placed into one of the sizes of the apparel (S, M, L, or XL)
* Have had no recent abdominal/leg surgery
* Are physically able to apply and remove low-compression apparel safely

Exclusion Criteria:

* Those on any special diets/medications that may affect weight especially hormone treatments that are changing such as IVF cycles
* Any malignancy that is being actively investigated or treated
* Any medical condition that is being actively investigated or treated
* Anyone who is on special diets for weight loss or other health issues, with the exception of those on stable diets such a gluten free for coeliac.
* Previous DVT
* (Unusual/abnormal) leg swelling
* Those who have had abdominal/leg operations within 1 year
* Those who are not mobile
* Those who are pregnant or planning to get pregnant

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This is based on sex not gender.
Enrollment: 24 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-04-03 (Estimated); Study Completion 2023-04-03 (Estimated)

PRIMARY OUTCOMES:
To calculate the volume of dimpling from the 3D scanner | 9 weeks
  Use this to objectively determine whether there is a change in appearance of cellulite with compression

SECONDARY OUTCOMES:
Using a visual analogue score for the participants and two blinded observers to score the appearance of cellulite from 0 to 10, 0 being the worst, 10 being the best to statistically analyse whether the opinion of cellulite has changed | 9 weeks
  Allows for statistical analysis between scores to see if there is a significant difference between the two.

CONTACTS AND LOCATIONS:
Locations (1):
- The Whiteley Clinic, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Derived] Kiely MJ, Poulsen A, Muschamp SD, Sallis C, Whiteley MS. Participant Reported Improvement in Cellulite by Vari-Pad Apparel and Objective Measurements - A "First Use" Pilot Study. Clin Cosmet Investig Dermatol. 2023 Sep 20;16:2573-2583. doi: 10.2147/CCID.S426978. eCollection 2023. PMID 37750084